CLINICAL TRIAL: NCT03305926
Title: Connected Rehabilitation: an Alternative to Conventional Cardiovascular Rehabilitation? Randomised Controlled Non-inferiority Trial in Patients With Coronary Artery Disease
Brief Title: Connected Rehabilitation: an Alternative to Conventional Cardiovascular Rehabilitation?
Acronym: eRCV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to changes in care management following the COVID context (remote/connected rehabilitation)
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASILLAS FRM 2016
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional CVR (Active Comparator)
  Interventions: Other: Conventional CVR programme; Other: Follow-up visit M2; Other: Follow-up vsit M8
- eCVR (Experimental)
  Interventions: Other: Connected CVR programme; Other: Follow-up visit M2; Other: Follow-up vsit M8

INTERVENTIONS:
Other: Conventional CVR programme — Programme in a CVR centre involving 20 sessions of reconditioning to effort, 3 times per week for roughly 7 weeks, as well as 14 sessions of therapeutic education in groups.
  Arms: Conventional CVR
Other: Connected CVR programme — First week in the CVR centre with 3 sessions combining reconditioning to effort, individual interviews and targeted therapeutic education, so as to define the objectives and methods of the connected CVR at home for the 6 following weeks.
  Arms: eCVR
Other: Follow-up visit M2 — Effort test and evaluation at the end of the CVR programme
Other: Follow-up vsit M8 — Evaluation at 8 months following the CVR programme

SUMMARY:
Cardiovascular rehabilitation (CVR) has major beneficial effects by improving physical capacity, accelerating return to activities and reinsertion and reducing mortality. It associates reconditioning to effort and therapeutic education for the optimal control of " risk factors ". It corresponds to a global approach to patients, thus counterbalancing the tendency to hyperspecialise in medicine. However, because of the lack of specialised centres, only a small proportion of patients (≈30%) are able to benefit. Numerical tools used in e-health, the deployment of the Internet and certain " connected " devices may provide alternatives outside hospital, by enabling the follow-up of patients and their physiological parameters (heart rate, blood pressure, weigh, physical activity…), and the adaptation - using an interactive web platform - of the physical activity programme, nutrition, compliance with medication and weaning from smoking. This project proposes to evaluate the effects of a so-called " connected " CVR programme, and to show its non-inferiority compared with a conventional CVR.

ELIGIBILITY:
Inclusion Criteria:

* men or women,
* aged between 30 and 75 years,
* presenting coronary artery disease without heart failure (Left ventricular ejection fraction on echocardiography (Simpson method) > 45 %).
* Patients who have provided written consent.

Exclusion Criteria:

* Adults under guardianship
* Patients without national health insurance cover
* Pregnant or breastfeeding women
* Inability to use connected numeric devices even simple operations (tablette, cardiofrequency meter, BP monitor…)
* Heart failure, with a low or preserved left ventricular ejection fraction
* Contra-indication for cardiovascular rehabilitation :

  * Severe obstructive heart disease (severe and asymptomatic obstacle to left ventricular ejection)
  * Acute unstable coronary syndrome
  * Tight aortic valve stenosis
  * Severe progressive cardiac rhythm or conduction disorders without pacing and discovered during the initial stress test
  * Intracavitary thrombus
  * Presence of moderate to severe pericardial effusion
  * Severe pulmonary artery hypertension (systolic PAP >70mmHg)
  * Recent history of venous thromboembolism (previous 3 months)
  * Progressive inflammatory or infectious disease
  * Inability to engage in physical exercise
* Impaired executive functions making it impossible to understand and comply with the CVR programme (Mini Mental Test < 24)
* Heart transplant
* Associated medical condition likely to impair functional capacities (examples: non-stabilised metabolic disorders such as progressive kidney failure, severe asthenia related to a severe non-stabilised disorder such as neoplasm, systemic diseases…)
* Physical disability in the lower limbs that could hamper reconditioning, whether neurological (central or peripheral), arterial (in particular, peripheral artery disease with a systolic index < 0.6) or orthopaedic (degenerative or inflammatory rheumatism)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
peak VO2, measured during an effort test | Month 2

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France